CLINICAL TRIAL: NCT01635179
Title: Laryngeal View With Intubation by Videolaryngoscopy With and Without Sellicks Maneuver.
Brief Title: Laryngeal View With Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Bjorn Arenkiel, Principal investigator, Glostrup University Hospital, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Glo-anaest-2012
Record Dates: First submitted 2012-06-19; First posted 2012-07-09 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Respiratory Aspiration; Hypoxemia
Keywords: Videolaryngoscopy; Bronchial Aspiration; Hypoxia
MeSH Terms: conditions — Respiratory Aspiration; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cricoid pressure (Experimental): A cricoid pressure of 30 N is done to occlude esophagus under a rapid sequence induction.
  Interventions: Procedure: Cricoid pressure

INTERVENTIONS:
Procedure: Cricoid pressure — The patient is intubated twice, once with a cricoid pressure and once with a sham-pressure, when performing a videolaryngoscopy.
  Other Names: Sellicks maneuver.; Profylaxis of bronchial aspiration

SUMMARY:
To prevent bronchial aspiration during induction of anaesthesia it has been a common procedure to perform a cricoid pressure, called Sellicks Maneuver, to occlude esophagus, and thereby prevent aspiration. During the last ten years the efficiency of this maneuver has been discussed, since it probably prolong the intubation time and do not significantly reduces the risk of aspiration.

The hypothesis is that Sellicks Maneuver prolong the time of intubation and reduces the view of the laryngeal inlet, during intubation with a videolaryngoscopy.

The hypothesis is tested by a double-blinded randomized study where patients is intubated twice, with and without Sellicks Maneuver, in a randomized order. The specific cricoid pressure is blinded to the personal performing the intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2, BMI < 35,
* no indication for rapid sequence induction,
* age > 18,
* able to give consent.

Exclusion Criteria:

* ASA > 2,
* BMI > 35,
* RSI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Completed intubation within 120 seconds | 120 seconds
  The primary outcome measure is the rate of completed and failed intubations. A intubations is failed when the oxygen saturation is less then 95% or the intubation time is longer then 120 seconds.

SECONDARY OUTCOMES:
A description of the laryngeal inlet | 120 seconds
  The secondary outcome measure is a description of the laryngeal inlet according the the Cormack-Lehan system, and how Sellicks Maneuver alters that view.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Arenkiel, MD, Principal Investigator — GlustrupUH dept of Anaesthesia
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark